CLINICAL TRIAL: NCT05887661
Title: The Application of Goal-directed Low Central Venous Pressure Based on Hypovolemic Phlebotomy in Laparoscopic Hepatectomy
Brief Title: Goal-directed LCVP Based on HP in Laparoscopic Hepatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shijiang Liu, MD, Clinical Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-SR-102
Record Dates: First submitted 2023-03-01; First posted 2023-06-05 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: hypovolemic phlebotomy; low central venous pressure; goal-directed; laparoscopic hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hypovolemic phlebotomy (HP) (Experimental): patients in this group undergoing laparoscopic hepatectomy was performed with goal-directed LCVP based on hypovolemic phlebotomy (HP)
  Interventions: Procedure: hypovolemic phlebotomy
- Control (No Intervention): patients in this group undergoing laparoscopic hepatectomy was performed with LCVP but no hypovolemic phlebotomy (HP)

INTERVENTIONS:
Procedure: hypovolemic phlebotomy — hypovolemic phlebotomy was performed after induction of anesthesia and before the star of parenchymal division, with a goal-directed low central venous pressure drop to 5mmHg.
  Other Names: HP
  Arms: hypovolemic phlebotomy (HP)

SUMMARY:
The goal of this clinical trial is to learn about goal-directed LCVP based on hypovolemic phlebotomy (HP) in laparoscopic hepatectomy. The main questions it aims to answer are:

1. The safety and feasibility of HP
2. To evaluate whether HP can reduce perioperative blood transfusion ratio Participants undergoing liver resection with HP was performed by the anesthesiologist. Blood was withdrawn approximately 30 min prior to the initiation of liver parenchymal transection from central venous. The aim was to maintain the CVP between 0 to 5 cmH2O. HP volume was 5-10 mL/kg of patient body weight, generally. Participants in control group undergoing liver resection without HP.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Hepatocellular Carcinoma
* Preference for laparoscopic hepatectomy and patient agreement

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Refusal of blood product transfusion
* Active cardiac conditions (unstable coronary syndromes, decompensated heart failure, significant arrhythmias, severe valvular disease, history of congestive heart failure)
* History of significant cerebrovascular disease
* Restrictive or obstructive pulmonary disease
* Uncontrolled hypertension
* Renal dysfunction (glomerular filtration rate <60 mL/min),
* Hemoglobin <100 g/L
* Abnormal coagulation values (international normalized ratio >1.5 not on warfarin and/or platelet count <100 ×109/L)
* Evidence of hepatic metabolic disorder (bilirubin >35 mmol/L)
* Presence of active infection
* Preoperative autologous blood donation
* Patients were not allowed to receive erythropoietin at any time during the index hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of allogeneic red blood cell products transfusion | From date of operation until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 12 months.
  The primary end point of the study was the proportion of patients who required transfusion of allogeneic red blood cell products during laparoscopic hepatectomy or at any time during the hospitalization during the index admission.

SECONDARY OUTCOMES:
The volume of Phlebotomy | From the start of operation until the end of operation.
The volume of Intraoperative blood loss | From the start of operation until the end of operation (during the operation).
The volume of Allogeneic transfusion (perioperative) | From date of operation until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 12 months.
The volume of Allogeneic transfusion (postoperative) | From the end of operation until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 12 months.
The volume of Allogeneic transfusion (intraoperative) | From the start of operation until the end of operation.
The volume of Fresh frozen plasm (FFP) transfusion | From date of operation until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 12 months.
The volume of Platelets transfusion | From date of operation until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 12 months.
The volume of Albumin transfusion | From date of operation until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 12 months.
Perioperative lowest concentration of Hb | From the start of operation until the date of discharge from hospital or date of death from any cause, whichever came first. assessed up to 12 months.
Pre-transection central venous pressure (CVP), (basic CVP) | From the start of anesthesia induction until the star of operation.
Lowest central venous pressure (CVP) | From the start of operation until the end of operation (during the operation).
time of pringle maneuver | From the start of operation until the end of operation.
number of pringle maneuver | From the start of operation until the end of operation.
  how many patients have the pringle maneuver
operating time | From the start of operation until the end of operation.
The proportion of laparoscopic hepatectomy converted to open liver resection | From the start of operation until the end of operation.
Length of stay | From date of hospitalization until the date of discharge from hospital or date of death from any cause, whichever came first. assessed up to 12 months
Number of Participants with postoperative complications (overall) | From date of operation until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 1 months.

CONTACTS AND LOCATIONS:
Overall Officials: Shijiang Liu, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided